CLINICAL TRIAL: NCT06560606
Title: UCAN CAN-DU: Canada-Netherlands Personalized Medicine Network in Childhood Arthritis and Rheumatic Disease
Acronym: UCAN CAN-DU
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Genome Canada (Other); Genome Alberta (Other); The Arthritis Society, Canada (Other); ReumaNederland (Unknown); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Alberta Children's Hospital (Other); Ontario Genomics (Unknown)
Responsible Party: Principal Investigator, Rae Yeung, Professor, Staff Physician and Senior Scientist, The Hospital for Sick Children
Other Study IDs: 1771
Record Dates: First submitted 2024-04-30; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — DNA, RNA, plasma, serum, cell
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1 - Biologic Basis of JIA: The objectives for this group are to help researchers look at childhood arthritis and determine which management approach is best for each individual child.
  To be eligible for this group:
  Participant must be ≤ 18 years of age at time of study enrollment. Participant is suspected to have JIA. Participant has not received any treatment other than non-steroidal anti-inflammatory drugs, such as acetaminophen.
- Cohort 2 - Start Biologics: The objectives for this group are to help researchers develop a tool to predict response to therapy.
  To be eligible for this group:
  Participant ≤ 18 years of age at time of study enrollment. Participant has been diagnosed with JIA and arthritis is active. Participant will be starting, re-starting or switching to a new biologic therapy.
- Cohort 3 - Stop Biologics: The objectives for this group are to help researchers develop a tool to predict who will remain in remission after discontinuing therapy.
  To be eligible for this group:
  Participant ≤ 18 years of age at time of study enrollment. Participant has been diagnosed with JIA and arthritis is inactive. Participant will be stopping or tapering biologic therapy.
- Cohort 4: Extreme Phenotypes: The objective for this group is new gene discovery and drug target identification.
  To be eligible for this group:
  There is high suspicion of genetic contribution. Participants are severely affected with difficult to control arthritis or systemic disease.
  There is unexplained systemic inflammation with arthritis/arthralgia as a part of manifestations

SUMMARY:
Childhood arthritis is a chronic disabling disease. New medications called biologic therapies are now available to treat arthritis that target key biologic molecules that cause inflammation. Biologic therapies, while very effective in treating arthritis in children, may have serious side effects including infections and potentially cancers, and are very expensive and doctors don't know, which one to choose for which child. The investigators will develop tests that enable them to learn about the biology of each child's arthritis and be able to predict when and which biologic therapy to start and when to stop.

DETAILED DESCRIPTION:
UCAN CAN-DU is a multicenter observational cohort study that will collect prospective data from children with arthritis. Biologic samples, clinical data and patient reported outcomes will be collected.

In addition, the study will also include a health economics component which will include a number of complementary approaches for quantifying and comparing benefits and risks that promote evidence-based, patient centered health care. This will address both the personal and societal economic burden of disease and include qualitative methods to inform the measurement of preferences, economic and simulation modelling to assess the value of biomarker testing. The socioeconomic impact of biomarker based treatment will be evaluated.

All clinical, biological and patient-derived data will be collected at an aggregation point housed and managed by High Performance Computing 4 Health (HPC4Health), a private hospital-only secure cloud-computing service within Compute Canada and physically located at SickKids/UHN. These databases and apps include biospecimen data and data collected through the eHealth platform. This will enable the study team to share and integrate data in near real-time into analytic models throughout the study course; hence providing a near real-time feedback from bench to bedside and vice versa.

The analysis of the cohorts will help define and confirm the biologic pathways predictive of disease course, treatment response and disease remission. This knowledge will then be used to develop a comprehensive clinical predictive tool to guide effective and safe treatment of childhood arthritis.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1: - Biologic Basis of JIA

* ≤18 years*
* Active objective arthritis suspected to be JIA or diagnosed with JIA within 6 months of enrolment
* Treatment naïve except for NSAIDs, allowed to have received NSAIDS within 6 months of diagnosis

Cohort 2 - Start Biologics

* JIA diagnosis as per ILAR criteria (all subtypes)
* ≤18 years*
* Active arthritis
* For sJIA, active disease not necessarily with arthritis.
* Time of start, restart or switch biologic therapy: e.g. failure, insufficient/partial response or intolerance

Cohort 3 - Stop Biologics

* JIA diagnosis as per ILAR criteria (all subtypes)
* ≤18 years*
* Inactive disease
* Discontinuing/tapering biologics for inactive disease

Cohort 4: Extreme Phenotypes

* Unexplained systemic inflammation with arthritis/arthralgia as a part of manifestations
* High suspicion of genetic contribution
* Severely affected patients with difficult to control disease (ie failure of multiple biologics)

Exclusion Criteria:

Cohort 1 :

* Arthritis explained by another diagnosis
* Joint injections as previous treatment less than 4 weeks prior to enrollment

Cohort 2:

* Arthritis explained by any other cause
* Start on biologics as an indication for uveitis only

Cohort 3:

- Tapering scheme > 12 months to complete biologics stop

Cohort 4:

- Arthritis explained by another diagnosis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be recruited from the patient population of a UCAN study site.
Sampling Method: Non-Probability Sample
Enrollment: 4100 (Estimated)
Dates: Start 2018-08-24 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Prospectively collect essential clinical data elements from children with new onset JIA | Up to 24 months
Evaluate clinical outcomes associated with the use of therapeutic agents in children with JIA | Up to 24 months
Evaluate clinical outcomes associated with the de-prescribing of therapeutic agents in children with JIA | Up to 24 months
Prospectively collect essential clinical data elements from children with extreme phenotypes of JIA. | Up to 12 months
Prospectively collect essential biological data elements from children with new onset JIA | Up to 24 months
Evaluate biological outcomes associated with the use of therapeutic agents in children with JIA | Up to 24 months
Evaluate biological outcomes associated with the de-prescribing of therapeutic agents in children with JIA | Up to 24 months
Prospectively collect essential biological data elements from children with extreme phenotypes of JIA | Up to 12 months
Prospectively collect essential socioeconomic data elements from children with new onset JIA | Up to 12 months
Evaluate the socioeconomic impact associated with the use of therapeutic agents in children with JIA | Up to 12 months
Evaluate the socioeconomic impact associated with the de-prescribing of therapeutic agents in children with JIA | Up to 24 months
Prospectively collect essential socioeconomic data elements from children with extreme phenotypes of JIA | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rae SM Yeung, MD, PhD, FRCPC, Principal Investigator — The Hospital for Sick Children (SickKids), University of Toronto; Nico Wulffraat, MD, PhD, Principal Investigator — Wilhelmina Children's Hospital, University Medical Center Utrecht; Susa Benseler, MD, PhD, Principal Investigator — Alberta Children's Hospital and Cumming School of Medicine, University of Calgary; Joost Swart, MD, PhD, Principal Investigator — Wilhelmina Children's Hospital, University Medical Center Utrecht; Bas Vastert, MD, PhD, Principal Investigator — Wilhelmina Children's Hospital, University Medical Center Utrecht
Locations (19):
- Canada (12):
  - Alberta Children's Hospital - University of Calgary, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Children's Hospital Health Science Centre Winnipeg, Winnipeg, Manitoba
  - Janeway Children's Hospital and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital, London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Montréal Children's Hospital, Montreal, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan
- Netherlands (7):
  - Amalia Children's Hospital, Radboudumc, Nijmegen, Gelderland
  - Sint Maartenskinderkliniek, Boxmeer, North Brabant
  - Emma Children's Hospital, Amsterdam UMC, Amsterdam, North Holland
  - Willem-Alexander Children's Hospital, LUMC, Leiden, South Holland
  - Sophia Children's Hospital, EMC, Rotterdam, South Holland
  - Beatrix Children's Hospital, UMCG, Groningen
  - Wilhelmina Children's Hospital, UMCU, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Data Access Advisory Committee (DAAC) has been formed. The DAAC is an advisory body tasked with guiding, developing and implementing principals for data sharing and policy for data access, including development of subcommittees to be formed to review request for secondary analysis or secondary or ancillary projects. The DAAC reports to the Executive Committee.
  IPD will only be shared at the summary level and de-identified.
Supporting Information: Study Protocol, CSR
Time Frame: Data sharing requests will continuously be reviewed on a case-to-case basis. Time frames will be according to the most DAAC terms of reference and governance rules.
Access Criteria: The DAAC will review the requests for access to clinical data and biologic data/samples collected through the UCAN CAN-DU project for the purposes of addressing secondary research questions. Assessments include, but not limited to, scientific merits, research environment, potential impact and significance, feasibility, overlap with other research questions, financial plan, and involvement with patient partners.